CLINICAL TRIAL: NCT03031574
Title: A Phase 1, Single-Center, Single-Dose, 2-Way Crossover, Randomized Food-Effect and Non-Randomized Gender- and Age- Effect Pharmacokinetic Study of SUVN-D4010 Orally Administered in Healthy Subjects
Brief Title: A Study to Investigate the Effect of Food, Gender, and Age on the Pharmacokinetic Profile of SUVN-D4010 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Suven Life Sciences Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTP1S240105HT4
Record Dates: First submitted 2017-01-23; First posted 2017-01-25 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Cognitive Disorder
Keywords: Serotonin 4 (5-HT4) receptor; Phase 1
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Food Effect (Active Comparator): SUVN-D4010 tablets single dose
  Interventions: Drug: SUVN-D4010
- Gender Effect (Active Comparator): SUVN-D4010 tablets single dose
  Interventions: Drug: SUVN-D4010
- Age Effect (Active Comparator): SUVN-D4010 tablets single dose
  Interventions: Drug: SUVN-D4010

INTERVENTIONS:
Drug: SUVN-D4010 — Tablets

SUMMARY:
The purpose of the study is to evaluate the effect of food, gender, and age on the single-dose pharmacokinetics (PK) of SUVN-D4010.

DETAILED DESCRIPTION:
The main objective of the study is to evaluate the safety and tolerability of orally administered SUVN-D4010 under single-dose conditions in healthy adult male and female subjects and healthy elderly male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects, aged 18 to 45 years, inclusive; healthy female subjects, aged 18 to 45 years, inclusive; healthy elderly male subjects, aged ≥65 years.
* Have a body mass index (BMI) between 18.0 and 30.0kg/m2 (inclusive) and weigh at least 50 kg and no more than 100 kg.

Exclusion Criteria:

* History or presence of gastrointestinal, hepatic, or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* Any clinically important illness, medical/surgical procedure, or trauma within 4 weeks of the (first) administration of the study drug.
* Any positive result at Screening for serum hepatitis B surface antigen, hepatitis C virus antibody, and human immunodeficiency virus antibody.
* Plasma or blood product donation within 1 month of the (first) administration of the study drug and any blood donation/blood loss more than 500 mL within the 2 months prior to the (first) administration of the study drug.
* As judged by the Investigator that the subject should not participate in the study if he/she is considered unlikely to comply with study procedures, restrictions, and requirements.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-01-23 (Actual); Primary Completion 2017-08-29 (Actual); Study Completion 2017-09-07 (Actual)

PRIMARY OUTCOMES:
Area under concentration (AUC) | 72 hours
Maximum observed concentration (Cmax) | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Dickerson, MD, PhD, Principal Investigator — PRA Health Sciences
Locations (1):
- PRA Health Sciences, Lenexa, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nirogi R, Bhyrapuneni G, Muddana NR, Goyal VK, Pandey SK, Mohammed AR, Ravula J, Jetta S, Palacharla VRC. First-in-Human Studies to Evaluate the Safety, Tolerability, and Pharmacokinetics of a Novel 5-HT4 Partial Agonist, SUVN-D4010, in Healthy Adult and Elderly Subjects. Clin Drug Investig. 2021 May;41(5):469-482. doi: 10.1007/s40261-021-01027-4. Epub 2021 Mar 31. PMID 33788154